CLINICAL TRIAL: NCT05503888
Title: An Open-label, Multicenter Phase Ib/II Clinical Study of Almonertinib Combined With SHR-1701 or Other Innovative Drugs in the Treatment of Relapsed or Advanced Non-small Cell Lung Cancer With EGFR Mutation
Brief Title: Phase Ib/II Study of Almonertinib Combined With SHR-1701 in the Treatment of Relapsed or Advanced Non-small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1701-215
Record Dates: First submitted 2022-08-08; First posted 2022-08-17 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Relapsed or Advanced Non-small Cell Lung Cancer
MeSH Terms: conditions — Recurrence | interventions — SHR-1701; aumolertinib

STUDY DESIGN:
Intervention Model Description: This study is a multicenter, open-label, dose-exploring, and efficacy expansion phase Ib/II study. The first phase explored two doses of SHR-1701 plus fixed dose of almonertinib to confirm RP2D. The second phase is for efficacy expansion through randomization.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Almonertinib combined with SHR-1701 (Experimental)
  Interventions: Drug: Almonertinib combined with SHR-1701
- Almonertinib (Placebo Comparator)
  Interventions: Drug: Almonertinib

INTERVENTIONS:
Drug: Almonertinib combined with SHR-1701 — Phase Ⅰb/Phase Ⅱ：
  SHR-1701: injection, intravenous infusion
  Almonertinib: tablets, oral
  Arms: Almonertinib combined with SHR-1701
Drug: Almonertinib — Phase Ⅱ:
  Almonertinib: tablets, oral
  Arms: Almonertinib

SUMMARY:
To evaluate the tolerability, safety, pharmacokinetic characteristics and immunogenicity of Almonertinib combined with SHR-1701 in relapsed or advanced NSCLC To evaluate the efficacy of Almonertinib combined with SHR-1701 in the first-line treatment of relapsed or advanced NSCLC

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily joined the study and signed informed consent
2. Age 18~75 years old, both male and female
3. Advanced NSCLC diagnosed by histology or cytology, or recurrent NSCLC after radical treatment such as surgery, radiotherapy, chemoradiotherapy
4. At least one measurable lesion based on RECIST v1.1 criteria
5. ECOG PS score: 0-1
6. Have a life expectancy of at least 3 months
7. Fertile women must have a negative serum pregnancy test within 3 days before the first dose and must be non-lactating

Exclusion Criteria:

1. Untreated Brain metastases with clinical symptoms; Or accompanied by meningeal metastasis, spinal cord compression，etc.
2. Uncontrolled pleural, pericardial, or abdominal effusion with clinical symptoms
3. Suffering from other malignant tumors in the past 3 years or at the same time
4. Presence of any active or known autoimmune disease
5. Subjects who had been systematically treated with corticosteroids (>10 mg/ day of prednisone or other equivalent hormone) or other immunosuppressive agents within 2 weeks prior to the first dose (randomization)
6. Any severe or uncontrolled ocular lesions that, in the judgment of the investigator, may increase the subject's safety risk
7. Have clinical symptoms or diseases of the heart that are not well controlled
8. Patients with hypertension who are not well controlled by antihypertensive medication
9. Any bleeding event of grade 2 or more or hemoptysis (volume of hemoptysis ≥2ml in a single episode) occurring within 2 weeks before the first dose (randomization); Clinically significant bleeding symptoms or definite bleeding tendency before the first medication (randomization)
10. Have known history of serious infections within 1 month prior to the first dose(randomization), including but not limited to infectious complications that require hospitalization, bacteremia, and severe pneumonia; use antibiotics within 1 week prior to the first dose(randomization); have any active infections requiring intravenous systemic therapy, or have a fever > 38.5°C of unknown cause before the first dose(randomization).
11. Have active or prior documented interstitial pneumonia/interstitial lung disease or pneumonitis that requires glucocorticoid treatment (e.g., radiation pneumonitis); Have active pneumonia at present
12. Have active pulmonary tuberculosis.
13. Have known history of human immunodeficiency virus (HIV) seropositive status or acquired immunodeficiency syndrome (AIDS). Have known active hepatitis B or C.
14. Had received lung radiation therapy within 6 months before the first dose (randomization); Had received major surgical treatment (except diagnostic surgery), systemic chemotherapy, immunotherapy, or other investigational drugs within 4 weeks prior to the first medication (randomization); Received palliative radiotherapy within 2 weeks before the first dose (randomization); Oral administration of molecular targeted drugs, less than 5 half-lives before discontinuation of the drug to the first dose (randomization); Failure to recover from toxicity and/or complications of previous interventions to NCI-CTC AE grade≤1

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity （Phase Ib） | 21 days after the first dose
The incidence and severity of ≥ grade 3 treatment-related adverse events (TRAE) and serious adverse events (TRSAE) in the combination of two drugs （Phase Ib） | from the time when all informed subjects signed the informed consent to the end of the safety follow-up period
PFS rate at 12 months | 12 months after the first medication for the last subject
  Progression-Free-Survival, defined as the time from randomization to the first occurrence of disease progression or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Adverse Events and Serious Adverse Events | up to 3 years
Proportion of dose pauses, dose downgrades and dose terminations due to study-drug related toxicities during the trial | up to 3 years
ORR | up to 3 years
DCR | up to 3 years
  Disease Control Rate, determined using RECIST v1.1 criteria
DoR | up to 3 years
  Duration of Response, determined using RECIST v1.1 criteria
DepOR | up to 3 years
  Depth of tumor remission, determined using RECIST v1.1 criteria
PFS | up to 3 years
  Progression-Free-Survival, determined using RECIST v1.1 criteria
OS | up to 5 years
  OS is the time interval from the date of randomization to death due to any reason or lost of follow-up

IPD SHARING:
Plan to Share IPD: Undecided